CLINICAL TRIAL: NCT02310867
Title: Immunomodulation to Optimize Vascularized Composite Allograft Integration for Limb Loss Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Linda Cendales (Other)
Responsible Party: Sponsor-Investigator, Linda Cendales, Associate Professor of Surgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00056079
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-02

CONDITIONS: Immunosuppression
Keywords: hand transplantation, amputation
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hand transplant with Belatacept (Experimental)
  Interventions: Drug: Belatacept; Procedure: Hand transplant

INTERVENTIONS:
Drug: Belatacept — This study will also test a new immunosuppressant drug called Nulojix® (belatacept) to see if it is able to prevent rejection in a hand transplant. Nulojix® (belatacept) is approved by the FDA for use in kidney transplants; however, it is investigational in this study.
  Other Names: Nulojix
Procedure: Hand transplant — The purpose of this study is to see if a surgical procedure for transplantation of a hand from a deceased donor can help subjects perform daily living activities better than they are currently able to do.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of hand transplantation as a treatment for patients with loss of limb below the elbow, The study will focus on patients who have had loss of limb. The primary endpoint is the ability to use the tranplanted limb in activities of daily living at 18 months following transplantation measured by a quantitative functional test.

Study activities include several study visits over 18 months and include; demographics, medical history, vital signs, psychosocial evaluation, urine, blood test, chest x-ray, bone density scans, and biopsies. Subjects who are 18-65 and willing to travel to site and have loss of limb will be included in study evaluation.

Risks of the study include risk of rejection and infection after being transplanted. Additional risk are associated with procedures that include blood draws, biopsies, x-rays, and potential loss of confidentiality. All patient data will be kept electronically and in accordance with the requirements of Duke University. In addition to the experimental data, this database includes recipient and donor demographics and transplant relevant medical history, range of motion, sensation, and immunosuppressive medications. Data will be recorded and reported in accordance with the standards required by the United Network for Organ Sharing (UNOS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients from 18-65 years old with loss of limb
2. Willingness and legal ability to give informed consent
3. Willingness to travel to study site for protocol specific samples to be taken, or in some cases, the ability to send samples via overnight mail

Exclusion Criteria:

* Any condition that precludes serial follow-up
* Any condition that would likely increase the risk of protocol participation or confound the interpretation of the data
* Any active malignancy or any history of a malignancy or lymphoma
* Inability or unwillingness to comply with protocol monitoring and therapy and immunodeficiency syndrome(s)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Ability to use the tranplanted limb in activities of daily living at 18 months following transplantation measured by a quantitative functional test. | 18 months

SECONDARY OUTCOMES:
Clinical rejection | 18 months
  Presence of macroscopic changes in the skin like a rash
Histological rejection | 18 months
  Presence of infiltrates categorized by the Banff classification

CONTACTS AND LOCATIONS:
Overall Officials: Linda Cendales, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States